CLINICAL TRIAL: NCT07277023
Title: The Influence of micro-and Macro Vascular Dysfunction on Clinical Severity in Adults With Sickle Cell Anemia (SS) and Sickle Cell Hemoglobin C Disease (SC)
Acronym: VASCUDREPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RBM-PAP-2015/108
Record Dates: First submitted 2017-11-27; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2017-11

CONDITIONS: Sickle Cell Anemia
Keywords: vascular dysfunction; sickle cell anemia; hemoglobin C disease
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobin C Disease

STUDY DESIGN:
Intervention Model Description: SCD patients are characterized by vascular alterations, with vascular function being severely affected. However, the exact contribution of vascular dysfunction in the clinical severity and the risk for frequent vaso-occlusive crises in SCD is unknown. Furthermore the factors involved in this imbalance remain unclear but it is supposed that cerebral hypoxia, the deficit in nitric oxide, abnormal blood rheology, increased microparticles levels, autonomic nervous system imbalance and a low level of physical activity as well as poor physical fitness might be involved.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- functions micro and macro-vascular in connection the clinical (Other): To characterize the level of alteration of micro and macro vascular function in SCD (SS, SC and Sß°) adults measured by heat-mediated vasodilation and peripheral perfusion (Laser Doppler system) and pulse wave velocity and to test relationships between this measured vascular function and clinical severity which is based on the rate of vaso-occlusive crisis (severe if ≥ 3 per year), the rate of acute chest syndrome (severe if > 0 per year) and/or the presence of chronic complications.
  Interventions: Diagnostic Test: The influence of micro-and macro vascular dysfunction on clinical severity in adults with sickle cell anemia (SS) and sickle cell hemoglobin C disease (SC)

INTERVENTIONS:
Diagnostic Test: The influence of micro-and macro vascular dysfunction on clinical severity in adults with sickle cell anemia (SS) and sickle cell hemoglobin C disease (SC) — The study permit to characterize the level of alteration of micro and macro vascular function in SCD (SS, SC and Sß°) adults measured by heat-mediated vasodilation and peripheral perfusion (Laser Doppler system) and pulse wave velocity and to test relationships between this measured vascular function and clinical severity which is based on the rate of vaso-occlusive crisis (severe if ≥ 3 within the 2 preceding years) and the rate of acute chest syndrome (severe if > 0 in the last 2 years).

SUMMARY:
The primary aim of this study is to determine the implication of micro and macro vascular function on the clinical severity of SCD (SS, SC, Sß°) adults. The secondary aim of this study is to understand the contribution of several parameters, known to influence vascular function in non-SCD individuals, in SCD

DETAILED DESCRIPTION:
TSCD patients are characterized by vascular alterations, with vascular function being severely affected. However, the exact contribution of vascular dysfunction in the clinical severity and the risk for frequent vaso-occlusive crises in SCD is unknown. Furthermore the factors involved in this imbalance remain unclear but it is supposed that cerebral hypoxia, the deficit in nitric oxide, abnormal blood rheology, increased microparticles levels, autonomic nervous system imbalance and a low level of physical activity as well as poor physical fitness might be involved.

* Primary outcome: The primary outcome of the present study is to characterize the level of alteration of micro and macro vascular function in SCD (SS, SC and Sß°) adults measured by heat-mediated vasodilation and peripheral perfusion (Laser Doppler system) and pulse wave velocity and to test relationships between this measured vascular function and clinical severity which is based on the rate of vaso-occlusive crisis (severe if ≥ 3 per year), the rate of acute chest syndrome (severe if > 0 per year) and/or the presence of chronic complications.
* Secondary outcomes: To test the existence of relationships between several factors: biological (hematology, blood rheology, nitric oxide and microparticles), physiological (the autonomic nervous system activity measured by Holter electrocardiogram and tissue oxygenation (muscular and cerebral)) and physical activity level (estimated by questionnaire and accelerometer) and physical fitness (estimated by the six minute walk test with oxygen consumption measurements).
* Study design: This study has been designed as biomedical, monocentric prospective and interventional study

ELIGIBILITY:
Inclusion Criteria:

* adults ≥ 18 years old,
* medical diagnosed with SCD (genotype SS, SC or Sß°) by isoelectrofocusing or HPLC at clinical steady state at the time of the study (i.e., no blood transfusion within the last three months,
* absence of acute episodes of infection, vaso-occlusive crisis or acute chest syndrome at least one month before inclusion in the study),
* regularly followed by the Sickle Cell Unit of the Academic Hospital of Pointe-à-Pitre (Guadeloupe) and having signed well informed the letter of agreement.

Exclusion Criteria:

* not at "steady-state";
* pregnancy or breast feeding;
* non-compliant patients to usual care;
* no signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-04-29 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Microvascular Function | Through study completion, an average of 3 years
  What is measured: Peripheral microvascular function will be assessed using Laser Doppler flowmetry to measure hyperemia response induced by localized heat.
  Units: Perfusion units (PU)
Macrovascular Function (Arterial Stiffness) | Assessed through study completion, average follow-up 3 years
  What is measured: Arterial rigidity will be evaluated using pulse wave velocity (PWV) measurements.
  Units: meters/second (m/s)

SECONDARY OUTCOMES:
Hematological and Hemorheological Profile Complete blood count | Through study completion, an average of 3 years
  Units: g/dL (hemoglobin),
Oxidative Stress Profile | Through study completion, average follow-up 3 years
  Plasma and erythrocyte markers of oxidative stress (e.g., malondialdehyde, glutathione).
  Units: μmol/L or standardized assay units
Circulating Nitric Oxide Levels | Through study completion, average follow-up 3 years
  Plasma concentration of nitric oxide metabolites. Units: μmol/L
Circulating Microparticles | Through study completion, average follow-up 3 years
  Number and origin of circulating microparticles (platelet, leukocyte, erythrocyte, endothelial). Units: particles/μL
Autonomic Nervous System Activity | Through study completion, average follow-up 3 years
  Heart rate variability (HRV) derived from Holter ECG recordings. Units: ms (standard deviation of NN intervals), normalized units (frequency domain parameters)
Muscle and Cerebral Oxygenation | Through study completion, average follow-up 3 years
  Oxygen saturation of muscle and brain tissue using near-infrared spectroscopy (NIRS). Units: % oxygen saturation
Physical Activity and Capacity 6-minute walk test distance | Through study completion, average follow-up 3 years
  Units: meters (walk test),
Effect of Hydroxyurea on Vascular Function | Through study completion, average follow-up 3 years
  Units: Perfusion units (microvascular), m/s (pulse wave velocity)
Hematological and Hemorheological Profile hematocrit | Thought study completion , an average of 3 years
  Units: % (hematocrit),
Hematological and Hemorheological Profile blood viscosity parameters | Through study completion, an average of 3 years
  mPa·s (blood viscosity)
Physical Activity and Capacity oxygen consumption (VO2) | Through study completion, average follow-up 3 years
  mL/kg/min (VO2)
Physical Activity and Capacity Accelerometer | Through study completion, average follow-up 3 years
  activity counts

CONTACTS AND LOCATIONS:
Overall Officials: Marie BILLAUD, Doctor in the Sickle Cell, Principal Investigator — Hospital University Center of Pointe-à-Pitre
Locations (1):
- Hospital University Center of Pointe-à-Pitre, Pointe-à-Pitre, Guadeloupe, Guadeloupe

IPD SHARING:
Plan to Share IPD: No